CLINICAL TRIAL: NCT05498155
Title: A Phase II, Multicentre, Open-Label Study to Assess the Efficacy and Safety of Olaparib Monotherapy and Olaparib Plus Durvalumab Combination as Neoadjuvant Therapy in Patients With BRCA Mutations and Early Stage HER2-Negative Breast Cancer
Brief Title: Study of Neoadjuvant Olaparib Monotherapy and Olaparib and Durvalumab Combination in HER2 Negative BRCAm Breast Cancer
Acronym: OlympiaN
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D931CC00001; 2023-503529-20-00 (Registry Identifier: CTIS (EU)); 2021-005231-22 (EudraCT Number)
Record Dates: First submitted 2022-07-05; First posted 2022-08-11 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer
Keywords: BRCA Mutations; Early Stage; HER2-Negative Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — olaparib; durvalumab

STUDY DESIGN:
Intervention Model Description: There will be 2 cohorts:
  Cohort A will consist of a lower-risk population Cohort B will consist of a higher-risk population Participants will be allocated to receive 300 mg oral olaparib twice daily as monotherapy or in combination with durvalumab 1500 mg via intravenous infusion every 4 weeks for a minimum of 4 and a maximum of six 28-day cycles before undergoing definitive surgery. Each participant will undergo definitive surgery, preferably within 6 weeks after receiving the final dose of neoadjuvant olaparib therapy, followed by standard treatment (radiation therapy, systemic therapy per institutional standards). Participants who achieve pCR at surgery, will be allowed to continue on treatment with olaparib in the adjuvant setting in lieu of standard adjuvant systemic therapy, per physician's choice. If the physician chooses adjuvant olaparib, then the total duration of olaparib therapy in the neoadjuvant and adjuvant setting should be 12 cycles.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort A (Experimental): Cohort A will consist of a lower-risk population of participants with HER2-negative ER-negative or ER-low defined as having a tumour size >5 mm and ≤20 mm and N0 (T1b-c/N0).
  Interventions: Drug: Neoadjuvant Olaparib monotherapy group
- Cohort B (Experimental): Cohort B will consist of a higher-risk population of participants with HER2-negative ER-negative or ER-low defined as having a tumour size of >20 mm but ≤50 mm and N0 (T2/N0), or having a tumour size of >1 mm but ≤20 mm and N1 (T1/N1).
  Interventions: Combination Product: Neoadjuvant combination therapy with olaparib plus durvalumab

INTERVENTIONS:
Drug: Neoadjuvant Olaparib monotherapy group — Neoadjuvant olaparib monotherapy (300 mg BID) for four to six 28-day cycles.
  Other Names: Cohort A
  Arms: Cohort A
Combination Product: Neoadjuvant combination therapy with olaparib plus durvalumab — Neoadjuvant combination therapy with olaparib (300 mg BID) plus durvalumab (1500 mg IV Q4W) for four to six 28-day cycles.
  Other Names: Cohort B
  Arms: Cohort B

SUMMARY:
This study to learn more about olaparib and olaparib plus durvalumab combination therapy and also to better understand the studied disease, breast cancer, and associated health problems.

Olaparib is a type of drug called a PARP (poly [adenosine diphosphate-ribose] polymerase) inhibitor. PARP inhibitors can destroy cancer cells that are not good at repairing DNA damage. Olaparib is also approved by US Food and Drug Administration (FDA), European Medicines Agency (EMA) and in other countries for treating women with BRCA-mutated, human epidermal growth factor receptor 2 (HER2)-negative metastatic breast cancer.

Durvalumab is a type of anticancer drug called immunotherapy that targets cancer cells by blocking the signal that prevents the immune system from seeing the cancer cell. Your immune system can then attack and kill the cancer cells. Durvalumab is approved by the FDA and the EMA for the treatment of patients with locally advanced non-small cell lung cancer after receiving chemoradiation therapy and extensive-stage small cell lung cancer in combination with chemotherapy.

Some parts of this study are experimental, which means that durvalumab and the combination of olaparib and durvalumab are still in the development stage for the treatment of breast cancer, and they are not approved for treatment of breast cancer, except for use in research studies like this.

DETAILED DESCRIPTION:
The investigation of olaparib as monotherapy or olaparib in combination with durvalumab in patients with early stage BRCAm, oestrogen receptor (ER)-negative or ER-low, human epidermal growth factor receptor 2 (HER2)-negative breast cancer who are candidates for neoadjuvant therapy supports the ongoing effort to identify novel agents and new drug combinations that can improve pathological complete response (pCR) rates and event-free survival (EFS). In patients at a lower risk (T1b-c/N0) of disease recurrence and a higher chance for cure, monotherapy olaparib may provide adequate neoadjuvant treatment. In contrast, monotherapy olaparib may be inadequate neoadjuvant treatment for those patients at a higher risk (T2/N0 or T1/N1) of recurrence, and the addition of an immune checkpoint inhibitor (ICI) to the neoadjuvant regimen may improve long-term outcomes as was seen in KEYNOTE-522 and GeparNuevo. However, the risk of irreversible immune-mediated adverse events (AEs) of the endocrine system due to ICI use supports the use of ICIs only in the cohort of patients at higher risk for disease recurrence. For both the lower and higher risk groups, the study treatments have the potential for the development of de-escalation strategies in this disease setting where traditional chemotherapy regimens may be avoided altogether.

While assessment of the efficacy of the combination of olaparib and durvalumab is ongoing, there are sufficient safety data available to develop a safety and tolerability profile for the combination.

ELIGIBILITY:
Inclusion Criteria:

* Males or Females ≥18 years
* Minimum body weight of 30 kg
* Capable of giving signed informed consent.
* Male and Female participants of childbearing potential must use effective methods of contraception
* Histologically confirmed, newly diagnosed, primary, operable, nonmetastatic invasive breast cancer with the following characteristics:

  --ER-negative or ER-low defined as IHC nuclear staining ≤10%
* HER2-negative (not eligible for anti-HER2 therapy) defined as:

  * IHC 0, 1+ without in situ hybridization OR
  * In situ hybridization non-amplified with ratio less than 2.0 OR
  * In situ hybridization average HER2 copy number < 6 signals/cells
* Clinical TNM staging (per AJCC 8th Edition) as follows:

  * T1b (>5 mm but ≤10 mm), N0, no known metastases (M0 or MX); OR
  * T1c (>10 mm but ≤20 mm), N0, no known metastases (M0 or MX); OR
  * T1 (>1 mm but ≤20 mm), N1, no known metastases (M0 or MX); OR
  * T2 (>20 mm but ≤50 mm), N0, no known metastases (M0 or MX).).
* Documented deleterious or suspected deleterious mutation in BRCA1 or BRCA2 from local BRCA testing using either a germline or tumour test.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Participants must have adequate organ and bone marrow function
* Participant must be willing to undergo a baseline research biopsy prior to start of study treatment.
* Participant must be willing to have any leftover tumour tissue/FFPE from the diagnostic biopsy submitted for research purposes, if available.

Exclusion Criteria:

* Any evidence of other diseases (such as severe or uncontrolled systemic diseases or active, uncontrolled infections, including but not limited to, uncontrolled ventricular arrhythmia, uncontrolled hypertension, recent [within 3 months] myocardial infarction, uncontrolled major seizure disorder, renal transplant, active bleeding diseases, unstable spinal cord compression, superior vena cava syndrome, extensive interstitial bilateral lung disease on High Resolution Computed Tomography scan
* Refractory nausea and vomiting, chronic gastrointestinal disease likely to interfere with absorption of the study medication, inability to swallow the formulated product
* History of another primary malignancy except for malignancy treated with curative intent with no known active disease for ≥5 years before the first dose of study intervention and of low potential risk for recurrence
* Participants with MDS or AML
* For higher risk (Cohort B) participants only: Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [eg, colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, sarcoidosis, granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc), autoimmune pneumonitis, and autoimmune myocarditis
* Known active hepatitis infection, positive hepatitis C antibody, hepatitis B virus surface antigen or hepatitis B virus core antibody
* Known to have tested positive for human immunodeficiency virus unless currently on effective anti-retroviral therapy with an undetectable viral load within 6 months
* History of arrhythmia (multifocal premature ventricular contractions, bigeminy, trigeminy, ventricular tachycardia), which is symptomatic or requires treatment (Common Terminology Criteria for Adverse Events [CTCAE] Grade 3), symptomatic or uncontrolled atrial fibrillation despite treatment, or asymptomatic sustained ventricular tachycardia
* Participant must not have had any prior treatment for the current breast cancer, including surgery, chemotherapy, hormonal therapy, radiation, or experimental therapy
* For higher risk (Cohort B) participants only: Prior exposure to anti-PD1, anti-PD-L1, or anti-CTLA4 agents (ICIs); OR an agent directed to other co-inhibitory or co-stimulatory T-cell receptors
* Any concurrent anticancer treatment
* Major surgical procedure (excluding placement of vascular access, local surgery of isolated lesions, or diagnostic staging) within 2 weeks of the first dose of study intervention
* For higher risk (Cohort B) participants only: Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab.
* Concomitant use of:

  * Known strong cytochrome P450 (CYP3A) inhibitors or moderate CYP3A inhibitors within 2 weeks prior to first dose of study intervention
  * Known strong CYP3A inducers or moderate CYP3A inducers .The required washout period prior to starting study therapy is 5 weeks for enzalutamide or phenobarbital and 3 weeks for other agents

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-11-07 (Actual); Primary Completion 2024-11-20 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy, measured by pCR (pathological complete response) rate, of olaparib monotherapy and olaparib plus durvalumab combination therapy, as assessed by central pathology review. | Approx. 4 to 6 months
  pCR is defined as ypT0/Tis ypN0 (ie, no invasive residual in breast and the axillary lymph nodes on evaluation of the complete resected breast specimen and all sampled regional lymph nodes) following completion of neoadjuvant systemic therapy.

SECONDARY OUTCOMES:
To evaluate the efficacy, measured by pCR rate, of olaparib monotherapy and olaparib plus durvalumab combination therapy as assessed by local pathology review | Approx. 4 to 6 months
  pCR is defined as ypT0/Tis ypN0 (ie, no invasive residual in breast and the axillary lymph nodes on evaluation of the complete resected breast specimen and all sampled regional lymph nodes) following completion of neoadjuvant systemic therapy.
To evaluate the efficacy, measured by RCB (residual cancer burden), of olaparib monotherapy and olaparib plus durvalumab combination therapy as assessed by central pathology review | Approx. 4 to 6 months
  RCB index value using 6 variables to categorize response in 1 of 4 classes: RCB 0 (pCR), I (minimal RCB), II (moderate RCB), and III (extensive RCB).
To evaluate the efficacy, measured by RCB, of olaparib monotherapy and olaparib plus durvalumab combination therapy as assessed by local pathology review | Approx. 4 to 6 months
  RCB index value using 6 variables to categorize response in 1 of 4 classes: RCB 0 (pCR), I (minimal RCB), II (moderate RCB), and III (extensive RCB).
To evaluate the efficacy of olaparib monotherapy and olaparib plus durvalumab combination therapy in terms of change from baseline tumour volume. Tumour volume will be assessed by local radiology review. | Approx. 4 to 6 months
  Percentage change in tumour volume from baseline after 3 cycles of treatment will be measured using MRI.
  Baseline is defined as the most recent measurement prior to the first administration of study intervention. Percent change from baseline is defined as: (Difference in value between post-baseline volume and baseline volume) divided by baseline volume and multiplied by 100.
To evaluate the efficacy of olaparib monotherapy and olaparib plus durvalumab combination therapy in terms of change from baseline tumour volume. Tumour volume will be assessed by local radiology review. | Approx. 4 to 6 months
  Percentage change in tumour volume from baseline after 6 cycles of treatment will be measured using MRI.
  Baseline is defined as the most recent measurement prior to the first administration of study intervention. Percent change from baseline is defined as: (Difference in value between post-baseline volume and baseline volume) divided by baseline volume and multiplied by 100.
To evaluate the efficacy of olaparib monotherapy and olaparib plus durvalumab combination therapy by assessment of EFS (event-free survival). | Approx. 3 years
  EFS is defined as time from the first dose of study intervention administration to any of the following events: progression of disease that precludes surgery, local or distant recurrence after surgery, second primary malignancy (breast or other invasive cancers), or death due to any cause.
Safety and tolerability profile of olaparib monotherapy and olaparib plus durvalumab combination therapy by assessment of advers events and seriuos advers events (AEs/SAEs) | Through study completion, around 15 months for single patient
  Graded according to the Common Terminology Criteria for Adverse Event (CTCAE) grade and changes in CTCAE grade
The number of participants with adverse events /serious adverse events of olaparib monotherapy and olaparib plus durvalumab combination therapy. | Through study completion, around 15 months for single patient
  Data will include clinical observations, ECG parameters, haematology / clinical chemistry, vital signs assessed as the number of participants with adverse events.
Safety and tolerability profile of olaparib monotherapy when given as adjuvant therapy to participants who achieve pCR by assessment of AEs/SAEs | Through study completion, around 15 months for single patient
  Graded according to the Common Terminology Criteria for Adverse Event (CTCAE) grade and changes in CTCAE grade
The number of participants with adverse events / serious adverse events of olaparib monotherapy when given as adjuvant therapy to participants who achieve pCR. | Through study completion, around 15 months for single patient
  Data will include clinical observations, ECG parameters, haematology / clinical chemistry, vital signs assessed as the number of participants with adverse events.
Systolic blood pressure (SBP), diastolic blood pressure (DBP) | Through study completion, around 15 months for single patient
  millimeter of mercury (mmHg)
Body Temperature | Through study completion, around 15 months for single patient
  Celsius (°C)
Pulse rate (heart rate) | Through study completion, around 15 months for single patient
  Beats per minute (BPM)
Weight | Through study completion, around 15 months for single patient
  Kilograms (kg)

CONTACTS AND LOCATIONS:
Overall Officials: Anitra Fielding, MBChB, Study Director — AstraZeneca
Locations (35):
- United States (5):
  - Research Site, Greeley, Colorado
  - Research Site, Loveland, Colorado
  - Research Site, Boston, Massachusetts
  - Research Site, Portland, Oregon
  - Research Site, Philadelphia, Pennsylvania
- Research Site, Melbourne, Australia
- Austria (2):
  - Research Site, Rankweil
  - Research Site, Salzburg
- Belgium (2):
  - Research Site, Brussels
  - Research Site, Liège
- Germany (7):
  - Research Site, Augsburg, by
  - Research Site, Cologne
  - Research Site, Essen
  - Research Site, Hamburg
  - Research Site, Hanover
  - Research Site, Heidelberg
  - Research Site, München
- Israel (4):
  - Research Site, Jerusalem
  - Research Site, Kfar Saba
  - Research Site, Ramat Gan
  - Research Site, Rehovot
- Italy (4):
  - Research Site, Bologna
  - Research Site, Meldola
  - Research Site, Modena
  - Research Site, Roma
- Spain (9):
  - Research Site, A Coruña
  - Research Site, Barcelona
  - Research Site, Cáceres
  - Research Site, Hospitalet deLlobregat
  - Research Site, Lleida
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Seville
  - Research Site, Valencia
- Research Site, Nottingham, United Kingdom